CLINICAL TRIAL: NCT01547286
Title: Redistribution of Pulmonary Perfusion During Bronchoconstriction in Asthma
Brief Title: Imaging Study of the Lungs During an Allergic Asthma Attack
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Robert Scott Harris, M.D., Assistant Professor of Medicine, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2007P002386; 1R01HL086717-01A2 (NIH)
Record Dates: First submitted 2012-02-15; First posted 2012-03-07 (Estimated); Results first posted 2017-04-25 (Actual); Last update posted 2017-11-22 (Actual); Status verified 2017-10

CONDITIONS: Asthma; Atopy
Keywords: Asthma; Allergen Challenge; Cat allergen; Dust mite allergen; Airway Hyper-responsiveness; Positron Emission Tomography - Computed Tomography; Nitrogen isotopes; Blood flow
MeSH Terms: conditions — Asthma; Respiratory Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Allergic asthmatic (Experimental)
  Interventions: Biological: Standardized Cat Allergen Extract and Standardized Dust Mite Allergen; Radiation: Computed Tomography imaging, functional Positron Emission Tomography imaging; Drug: Nebulized methacholine inhalation

INTERVENTIONS:
Biological: Standardized Cat Allergen Extract and Standardized Dust Mite Allergen — The route of administration will be topical application of the titrated allergen via nebulized droplets to the lungs. The starting dose of allergen will be 3 dose dilutions below the estimated provocative concentration of allergen that causes a 20% fall in Forced Expired Volume in 1 second delivered for 5 minutes at tidal breathing, followed by Forced Expired Volume in 1 second at 10-minute intervals until the lowest Forced Expired Volume in 1 second is established. If the percent of Forced Expired Volume in 1 second fall is < 20%, the next concentration is given, until the Forced Expired Volume in 1 second falls ≥ 20 percent. When this happens the Forced Expired Volume in 1 second will be followed at 10, 20, 30, 45, and 60 minutes, then hourly for 7 hours. The early asthmatic response is the maximum percent of Forced Expired Volume in 1 second fall between 0 and 3 hours and the late asthmatic response between 3 and 7 hours post allergen challenge.
  Other Names: •Reagents from Greer will be used:; •Standardized Cat Hair Extract; •Standardized mite extract-Dermatophagoides farinae; •Standardized mite extract-Dermatophagoides pteronyssinus
Radiation: Computed Tomography imaging, functional Positron Emission Tomography imaging — Physiology study using Computed Tomography and Positron Emission Tomography imaging with Nitrogen-13 saline as radiotracer; images obtained during the early and late phases after allergen challenge
Drug: Nebulized methacholine inhalation — Standard methacholine challenge performed once to determine the subject's dose that causes a 20% fall in Forced Expired Volume in 1 second from baseline.
  Other Names: MethaPharm Provocholine

SUMMARY:
Asthma is a disease of rapidly increasing incidence that already affects more than 17 million people in the United States alone. It has long been known that areas of severely reduced airflow occur in asthma and contribute significantly to the impairment of gas exchange in this disease. However, the extent to which local blood flow changes during an asthmatic attack is unclear. The purpose of this study is using Positron Emission Tomography - Computed Tomography imaging to evaluate how the blood flow changes in the lungs during an asthma attack induced by allergens.

DETAILED DESCRIPTION:
Asthma is a disease of rapidly increasing incidence that already affects more than 17 million people in the United States alone. It is of major importance to understand the mechanisms responsible for underlying mechanical and physiological changes that occur during asthma exacerbations. The effect of asthma on the pulmonary vasculature is virtually unknown. It has long been known that areas of severely reduced airflow occur in asthma and contribute significantly to the impairment of gas exchange in this disease. However, the extent to which local blood flow changes during an asthmatic attack is unclear. This proposal is designed to evaluate the relevance of potential mechanisms responsible for the blood flow defects seen in our Positron Emission Tomography studies of subjects with asthma and identify factors modifying that perfusion distribution. With this knowledge, it is hoped that a more focused basic research is motivated to understand the fundamental mechanisms behind these processes ultimately targeted to improved asthma therapy. Comparing these measures in healthy subjects and asthmatics patients may lead to methods to improve patient care.

ELIGIBILITY:
Inclusion Criteria:

* Mild asthma is defined in the National Institutes of Health 2002 guidelines for the Diagnosis and Management of Asthma. Briefly, people with mild asthma are defined as those with symptoms greater than 2 times a week but less than once per day with normal Forced Expired Volume in 1 second (> 80% predicted)
* Clinical history of allergic symptoms to cat or dust mite allergen and demonstrated skin reactivity
* Life-long absence of cigarette smoking (defined as a lifetime total of less than 5 pack-years); none in 5 years
* Willing and able to give informed consent
* Expressed the desire to participate in an interview with the principal investigator

Exclusion Criteria:

* Women of childbearing potential who are documented to be pregnant (based on blood testing) or who are nursing.
* The presence of spontaneous asthmatic episode or clinical evidence of upper respiratory tract infection within the previous 6 weeks.
* Participation in research study involving a drug or biologic during the 30 days prior to the study.
* Intolerance to albuterol, atropine, or lidocaine.
* Antihistamines within 7 days of the screening visit.
* Known exposure to agents that are associated with pulmonary disease (i.e. asbestos, silica).
* Presence of other known pulmonary disease, coronary disease, congestive heart failure, ventricular arrhythmias, history of a cerebrovascular accident, renal failure (or creatinine > 1.5, if known), history of anaphylaxis, cirrhosis or presence of a significant disease, which in the opinion of the principal investigator, would pose a significant risk for the subject or confound the results of the study.
* Use of systemic steroids, increased use of inhaled steroids, beta blockers and mono-amine oxidase inhibitors or a visit for an asthma exacerbation within

  1 month of the screening visit.
* A history of asthma-related respiratory failure requiring intubation.
* A history of hospitalization for asthma.
* Subjects with a high possibility of poor compliance with the study as judged by the principal investigator.
* History of contrast dye allergy.
* Unresponsive to bronchodilator agents.
* Quantitative skin prick test at or below a dilution level of standardized cat allergen extract of 1:2048 (4.88 bioequivalent allergy unit/ml)for subjects being challenged with cat allergen.
* Quantitative skin prick test at or below a dilution level of standardized mite allergen extract of 1:2048 (4.88 bioequivalent allergy unit/ml)for subjects being challenged with either mite allergen.
* Subjects who, by participating in one of these studies, will have a cumulative radiation dose exceeding the maximum yearly recommended dose for a research subject (50 milliSieverts).
* Previous participation in one of the protocols in this proposal.
* Contraindication to methacholine challenge testing (Forced Expired Volume in 1 second < 50% predicted or < 1L, heart attack or stroke in last 3 months, uncontrolled hypertension, or known aortic aneurysm).
* Body Mass Index > 32

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2012-05; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: R. Scott Harris, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited using an IRB approved advertisement from December 2012 - January 2013. Potential subjects completed two screening visits, during which the informed consent was obtained, clinical assessment, spirometry, methacholine challenge and allergic skin tests were performed. All screening visits took place at our pulmonary clinics.
Pre-assignment Details: This is a single group design study. Subjects were instructed to withhold their asthma and allergy medications before the screening and bronchial allergen challenge tests. The duration of the medication withholding depended on which medications they were using at that time.
Groups:
- Allergic Asthmatic: This is a single physiological group study where each subject served as their own control. All eligible subjects underwent a methacholine challenge test, clinical assessment and skin tests to ascertain the diagnosis of allergic asthma. Both methacholine and skin test results were used to determine the start dose of the bronchial allergen challenge test. CT and PET with Nitrogen-13 (13NN) saline as a radiotracer images were obtained during the early and late phases after allergen challenge.
Period: Overall Study
Arm/Group | Allergic Asthmatic
Started | 7
Completed | 5
Not Completed | 2
Not completed — Did not meet all eligibility criteria | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Population: 7 Subjects were enrolled and 5 subjects completed the study. Demographics and metacholine challenge test were obtained from all 7 subjects.
Groups:
- Allergic Asthmatic: Standardized Cat Allergen Extract and Standardized Dust Mite Allergen: The route of administration will be topical application of the titrated allergen via nebulized droplets to the lungs. The starting dose of allergen will be 3 dose dilutions below the estimated PC20-allergen delivered for 5 minutes at tidal breathing, followed by FEV1 at 10-minute intervals until the lowest FEV1 is established. If the %FEV1 fall is < 20%, the next concentration is given, until the FEV1 falls ≥ 20%. When this happens the FEV1 will be followed at 10, 20, 30, 45, and 60 minutes, then hourly for 7 hours. The early asthmatic response is the maximum %FEV1 fall between 0 and 3 hours and the late asthmatic response between 3 and 7 hours post allergen challenge.CT imaging, functional PET imaging: Physiology study using CT and PET imaging with Nitrogen-13 (13NN) saline as radiotracer; images obtained during the early and late phases after allergen challenge. Nebulized methacholine inhalation: Standard
Arm/Group | Allergic Asthmatic
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.7 (5.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change in the Ratio of Mean-normalized Perfusion Within Ventilation Defective Regions Relative to Outside
Description: Blood flow relative to the mean blood flow of the lung (mean normalized perfusion) inside areas that have reduced ventilation (Vdefs) relative to outside the Vdefs. Or, another way of writing this is: (Blood flow inside Vdefs/mean blood flow of the lung)/(Blood flow outside Vdefs/mean blood flow of the lung).
Time Frame: 3 hours after allergen administration
Measure: Mean (Standard Deviation); unit: percentage
Groups:
- Allergic Asthmatic: Standardized Cat Allergen Extract and Standardized Dust Mite Allergen: The route of administration will be topical application of the titrated allergen via nebulized droplets to the lungs. The starting dose of allergen will be 3 dose dilutions below the estimated PC20-allergen delivered for 5 minutes at tidal breathing, followed by FEV1 at 10-minute intervals until the lowest FEV1 is established. If the %FEV1 fall is < 20%, the next concentration is given, until the FEV1 falls ≥ 20%. When this happens the FEV1 will be followed at 10, 20, 30, 45, and 60 minutes, then hourly for 7 hours. The early asthmatic response is the maximum %FEV1 fall between 0 and 3 hours and the late asthmatic response between 3 and 7 hours post allergen challenge.
  CT imaging, functional PET imaging: Physiology study using CT and PET imaging with Nitrogen-13 (13NN) saline as radiotracer; images obtained during the early and late phases after allergen challenge Nebulized methacholine inhalation: Standard
Arm/Group | Allergic Asthmatic
Number analyzed (Participants) | 5
percentage | -17.8 (5.1)

2. Primary Outcome: Percentage Change in the Ratio of Mean-normalized Perfusion Within Ventilation Defective Regions Relative to Outside
Description: as for outcome 1
Time Frame: 7 hours after allergen administration
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Allergic Asthmatic
Number analyzed (Participants) | 5
percentage | -26.3 (9.8)

3. Secondary Outcome: Coefficient of Variation Squared of Perfusion
Description: Coefficient of variation squared of the perfusion in the imaged lung. This measures the overall heterogeneity of perfusion in the imaged lung.
Time Frame: 3 hours after allergen administration
Measure: Mean (Standard Deviation); unit: unitless
Groups:
- Allergic Asthmatic: All subjects were allergic asthmatics, each served as their own control. There was no comparator group.
Arm/Group | Allergic Asthmatic
Number analyzed (Participants) | 5
unitless | 0.11 (0.03)

4. Secondary Outcome: Coefficient of Variation Squared of Perfusion
Description: as for outcome 3
Time Frame: 7 hours after allergen administration
Measure: Mean (Standard Deviation); unit: unitless
Arm/Group | Allergic Asthmatic
Number analyzed (Participants) | 5
unitless | 0.15 (0.07)

ADVERSE EVENTS:
Time Frame: Subjects were monitored throughout the study and there were no adverse events.
Groups:
- Allergic Asthmatic: Standardized Cat Allergen Extract and Standardized Dust Mite Allergen: The route of administration will be topical application of the titrated allergen via nebulized droplets to the lungs. The starting dose of allergen will be 3 dose dilutions below the estimated PC20-allergen delivered for 5 minutes at tidal breathing, followed by FEV1 at 10-minute intervals until the lowest FEV1 is established. If the %FEV1 fall is < 20%, the next concentration is given, until the FEV1 falls ≥ 20%. When this happens the FEV1 will be followed at 10, 20, 30, 45, and 60 minutes, then hourly for 7 hours. The early asthmatic response is the maximum %FEV1 fall between 0 and 3 hours and the late asthmatic response between 3 and 7 hours post allergen challenge.
  CT imaging, functional PET imaging: Physiology study using CT and PET imaging with Nitrogen-13 (13NN) saline as radiotracer; images obtained during the early and late phases after allergen challenge
Arm/Group | Allergic Asthmatic
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No